CLINICAL TRIAL: NCT00244660
Title: Blood Pressure Reduction in Danish General Practice (BRIDGE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.504
Record Dates: First submitted 2005-10-20; First posted 2005-10-27 (Estimated); Last update posted 2008-01-21 (Estimated); Status verified 2008-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Educational Status

INTERVENTIONS:
Procedure: Frequent blood pressure measurements
Behavioral: Education

SUMMARY:
To investigate the effect on blood pressure (BP) control in hypertensive patients using a combination of frequent home - and 24-h ambulatory blood pressure measurement (ABPM) in a Danish general practice (GP) setting.

DETAILED DESCRIPTION:
Also the beneficial effect of optimal blood pressure (BP) control is well established, sub-optimal blood pressure control is still highly prevalent in the hypertensive population. The purpose of this study is to evaluate the effect of frequent home (HBPM)- and 24 hour (ABPM) blood pressure measurements to achieve BP control in patients with essential hypertension according to Danish Society of Hypertension Gudelines. The study will include 120 general practioners (GP) randomised to perform either usual BP control or intensive BP control. Before randomization, participating GPs will recruit each 10 patients to be followed over a period of 12 months. At baseline ABPM will be measured in all eligible patients. The result of the baseline ABPM will be blinded in the usual care group. Following this, usual care (control) physicians will perform BP control according to their usual standard. Physicians randomized to intensive care will control BP by the use of frequent HBPM and ABPM. According to a pre-specified scheme patients followed by intensive care physicians will measure HBP in the morning and in the evening at three consecutive days after 1, 2, 4, 8 and 10 months in the study. Patients will communicate the results of these measurements to the treating physician, who according to the result of the HBPM will decide what action to take. As a further aid, at 6 month patients in the intensive care group will have another APBM as part of the follow up to ensure 24 hour BP control. In both the usual- and intensive care group all treatment decisions is entirely up to the treating physician. No pre-specified treatment algorithm has to be followed and both non-pharmacological as well as any pharmacological tretment can be used to (optimize) BP control. Patients followed by intensive care will receive extended structured information about the importance of optimal BP control. As the primary endpoint is change in mean 24-hour ambulatory systolic and diastolic blood pressure patients in both groups will have a ABPM after 12 months. During the whole trial, participating physicians will keep a record of all measured BP (clinic BP, HBP and ABP), as well as all relevant blood- and urinary tests (lipids, glucose, albuminuria) taken during the study. Based on all available information, patients total risk score (Danish Society of Hypertension) will be calculated at baseline and after 12 months.

Study Hypothesis:

Blood pressure control according to the Danish Society of Hypertension Guidelines is better obtained by an intensive care regimen (frequent home- and ambulatory blood pressure measurement) compared to a usual care regimen (standard blood pressure control in Danish general practice).

Comparison(s):

Frequent home- and ambulatory blood pressure measurements versus standard care.

ELIGIBILITY:
Inclusion criteria: 18 years or more, informed consent obtained, essential hypertension, able to use a home blood pressure apparatus, can cooperate to ambulatory blood pressure measurement. Exclusion criteria: Pregnancy, hypertension secondary to another disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2005-11; Study Completion 2007-06

PRIMARY OUTCOMES:
Change in mean 24-hour (ambulatory) systolic and diastolic blood pressure after 12 months.

SECONDARY OUTCOMES:
Change in clinic and home sysolic and diastolic blood pressure after 12 months, change in systolic and diastolic blood pressure the last 6 hours of the dosing interval (morning blood pressure) and change in over all risk score after 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Denmark A/S
Locations (1):
- Frederiksberg Hospital, Frederiksberg F, Denmark

REFERENCES:
- [Derived] Klarskov P, Bang LE, Schultz-Larsen P, Gregers Petersen H, Benee Olsen D, Berg RMG, Abrahamsen H, Wiinberg N. Intensive versus conventional blood pressure monitoring in a general practice population. The Blood Pressure Reduction in Danish General Practice trial: a randomized controlled parallel group trial. Fam Pract. 2018 Jul 23;35(4):433-439. doi: 10.1093/fampra/cmx106. PMID 29351658